CLINICAL TRIAL: NCT04666337
Title: Fentanyl Versus Tramadol as Co-administrator to Bupivacaine in Ultrasound-guided Supraclavicular Brachial Plexus Blockade: Pons and Cons
Brief Title: Fentanyl Versus Tramadol as Co-administrator to Bupivacaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, huda fahmy, Assistant professor of Anesthesia and Intensive Care, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 337/2/19
Record Dates: First submitted 2020-12-01; First posted 2020-12-14 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Acquired Deformity of Elbow; Forearm; Hand; Wrist
Keywords: Supraclavicular Brachial Plexus Blockade; Fentanyl; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomization established using the computer-generated closed envelopes method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group B (bupivacaine group) (Active Comparator): patients received 20 ml bupivacaine 0.5% plus normal saline (2ml)
  Interventions: Procedure: ultrasound-guided supraclavicular brachial plexus blockade
- Group F (fentanyl group) (Active Comparator): patients received 20 ml bupivacaine 0.5% plus fentanyl (100µg-2 ml)
  Interventions: Procedure: ultrasound-guided supraclavicular brachial plexus blockade
- Group T (tramadol group) (Active Comparator): patients received 20 ml bupivacaine 0.5% plus tramadol (100mg-2 ml)
  Interventions: Procedure: ultrasound-guided supraclavicular brachial plexus blockade

INTERVENTIONS:
Procedure: ultrasound-guided supraclavicular brachial plexus blockade — Ultrasound-guided supraclavicular brachial plexus block was done using an ultrasound machine (Philips; Model: OTD020, AcBel Polytech Inc., Taiwan) with a 5-10 MHz linear probe. The brachial plexus and its relation to the surrounding structures were viewed while the patient was supine and the head turned 45° to the contralateral side. In the supraclavicular fossa, the probe was placed in the coronal plane to visualize the subclavian artery and the brachial plexus in a transverse sectional view. After skin sterilization and local anesthetic administration, an insulated needle was then introduced lateral to the ultrasound probe and parallel to the long axis of the probe. Once the needle penetrated the brachial plexus cluster, the local anesthetic mixture was injected incrementally after negative aspiration for blood or air just next to the artery, then the needle was repositioned to inject on the upper pole of the artery.

SUMMARY:
Supraclavicular brachial plexus approach is an alternative technique to general anesthesia resulting in a fast onset of a reliable blockage of the brachial plexus. The use of ultrasound for the performance of supraclavicular block has become the gold standard since it enables the clinician to deposit the local anesthetic close to the nerves in real-time that improves the success rate with a safety margin. Adjuvants are added to local anesthetic in Supraclavicular Brachial Plexus Blockade to improve the quality of nerve blocks and the duration of analgesia. It should be noted that no adjuvant has been approved by the Food and Drug Administration (FDA) for the prolongation of peripheral nerve blocks

DETAILED DESCRIPTION:
There are multiple controversies among the previous studies for the use of different opioids as adjuvants for brachial plexus blockade to improve various block characteristics. Moreover, limited studies estimate the pons and cons of tramadol versus fentanyl as co-administrator to bupivacaine in Ultrasound-guided Supraclavicular Brachial Plexus Blockade.

In our study, we aim to assess the utility of fentanyl versus tramadol as co-administrator to bupivacaine in ultrasound-guided supraclavicular brachial plexus blockade in upper limb surgeries in a prospective randomized controlled fashion. The primary outcome is to compare between the efficacy of tramadol versus fentanyl as adjuvants on the onset and duration of sensory and motor block and the secondary outcome is to compare between the efficacy of tramadol versus fentanyl as adjuvants on postoperative analgesia, time of the request to rescue analgesia, postoperative analgesic consumption, and complications.

The patients were aged between 18 and 60, both gender, and the American Society of Anesthesiologists (ASA) physical status I/II. However, patients who had bleeding disorders got opioid analgesics or monoamine oxidase inhibitors before surgery, had a history of seizures, respiratory or cardiac diseases, local infections at the site where needle for the block is to be inserted, pregnant woman and in whom the block effect was partial and required supplementary anesthesia were excluded from the study.

Patients were randomly allocated into three groups for ultrasound-guided supraclavicular brachial plexus block. Randomization was established using the computer-generated closed envelopes method.

Group B (bupivacaine group): patients received 20 ml bupivacaine 0.5% plus 2 ml normal saline Group F (fentanyl group): patients received 20 ml bupivacaine 0.5% plus fentanyl (1µg/kg-2 ml) Group T (tramadol group): patients received 20 ml bupivacaine 0.5% plus tramadol (1mg/kg-2 ml)

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I/II. scheduled for forearm or hand surgery

Exclusion Criteria:

* bleeding disorders
* patients who got opioid analgesics or monoamine oxidase inhibitors before surgery,
* history of seizures, respiratory or cardiac diseases
* local infections at the site where the needle for the block is to be inserted
* a pregnant woman
* the block effect was partial and required supplementary anesthesia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Onset time of sensory block in minutes | 40 minutes
  After the injection of the solution, every patient was checked for the onset of sensory blockade using goose soaked with iced normal saline by the following scale (three-point scale): Grade 0= perceived as normal sensation, Grade 1 = loss of cold sensation (analgesia), Grade 2= loss of sensation of touch (anesthesia).
onset time of motor blockade in minutes using the modified Bromage scale (Three-point scale) | 40 minutes
  the modified Bromage scale (Three-point scale): Grade 0: Normal motor function, Grade 1: Decreased motor strength with the ability to move the fingers only, Grade 2: Complete motor block with an inability to move the fingers.
Duration of sensory block in hours | 24 hours
  It's the time from sensory block onset to the time of restoration of sensation at the surgical site
Duration of motor block in hours | 24 hours
  It's the time from motor block onset to the restoration of global mobility in the hand and the wrist.

SECONDARY OUTCOMES:
Visual analog scale (VAS): the VAS consisted of a straight, vertical 10-cm line; the bottom point represented "no pain" = (0 cm) and the top "the worst pain you ever have" = (10 cm). | 24 hours
  Patients were asked to rate their pain intensity at 1, 2, 4, 6, 12, 18, and 24 h after the block
Postoperative first analgesic request time in hours | 24 hours
  was taken from the time of complete sensory block to the request to rescue analgesia when VAS > 4 cm.
Rescue analgesia in the form of 0.05 mg/kg morphine sulfate intravenously | 24 hours
  was given when VAS ≥ 4 cm
Mean blood pressure in mmHg | 24 hours
  was measured before the block (0 min) and at 5, 10, 15, 30 min then 1, 2, 3, 6, 12,18and 24 h after the block
heart rate in beats / minute | 24 hours
  was measured before the block (0 min) and at 5, 10, 15, 30 min then 1, 2, 3, 6, 12,18and 24 h after the block.
peripheral oxygen saturation | 24 hours
  was measured before the block (0 min) and at 5, 10, 15, 30 min then 1, 2, 3, 6, 12,18and 24 h after the block.

CONTACTS AND LOCATIONS:
Overall Officials: huda fahmy, ph D, Principal Investigator — Aswan University
Locations (1):
- Aswan University Hospital, Aswān, Egypt